CLINICAL TRIAL: NCT07327580
Title: The Effect of Watson Human Care Theory and Acceptance and Commitment Therapy-Based Counseling Program Applied to Parents of Pediatric Palliative Care Patients on Value-Based Life and Care Burden
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Esma Ceren ŞİŞGİNOĞLU, PhD Student, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 27702
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Palliative Care; Caregiver Burden; Acceptance and Commitment Therapy
Keywords: pediatric palliative care; caregiver burden; acceptance and commitment therapy
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this arm will receive counseling based on Watson's Theory of Human Caring and Acceptance and Commitment Therapy (ACT).
  Interventions: Behavioral: Counseling Program Based on Watson Human Care Theory and Acceptance and Commitment Therapy (ACT)
- Control Group (No Intervention): Participants in this arm will receive usual care only, without any additional intervention.

INTERVENTIONS:
Behavioral: Counseling Program Based on Watson Human Care Theory and Acceptance and Commitment Therapy (ACT) — The subject of this research is to examine the effect of Watson Human Care Theory and Acceptance and Commitment Therapy-based counseling program applied to parents of pediatric palliative care patients on value-oriented life and care burden.
  Arms: Intervention Group

SUMMARY:
This study aims to examine the effect of Watson Human Care Theory and Acceptance and Commitment Therapy-based counseling program applied to parents of pediatric palliative care patients on value-oriented living and care burden.

ELIGIBILITY:
Inclusion Criteria:

* Being the parent of a patient in need of pediatric palliative care at the hospital where the study will be conducted during the dates of the study,
* Being between the ages of 18-65,
* Agreeing to participate in the study,
* Having the ability to read, write and understand Turkish,
* The patient with pediatric palliative care has been provided care for at least 1 month.

Exclusion Criteria:

* Having previously received similar therapy or psychoeducation or being involved in ongoing training,
* Having received a psychiatric diagnosis,
* Having communication problems such as hearing and vision,
* Being a foreign national,
* Not being the biological mother or father of the patient in need of pediatric palliative care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
valued living | Baseline and immediately post-intervention.
  Valued living will be assessed using a validated self-report questionnaire measuring the extent to which individuals live in accordance with their personal values.

SECONDARY OUTCOMES:
caregiver burden | Baseline and immediately post-intervention.
  Caregiver burden will be assessed using a validated self-report scale evaluating the perceived physical, emotional, and social burden associated with caregiving.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No